CLINICAL TRIAL: NCT06950151
Title: Cross-sectional Study on the Early Detection of Chronic Kidney Disease
Brief Title: Early Detection of Chronic Kidney Disease
Acronym: DetERC-GARRAF
Status: Completed | Type: Observational
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Other Study IDs: CSAPG-72
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic Kidney Disease Group: Patients with chronic kidney disease and at least one referral criterion for nephrology teleconsultation.

SUMMARY:
This retrospective observational study aims to assess the proportion of patients who were appropriately referred from primary care to the nephrology teleconsultation service. The appropriateness of the referral will be determined by the time elapsed between the referral criteria being met and the date of the teleconsultation, as well as by the patient's treatment at the time of referral.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age
* Teleconsultation to nephrology from Primary Care in the Garraf region during the period from January to December 2024
* Patients with at least one referral criterion for the nephrology service

Exclusion Criteria:

Participants diagnosed with any of the following conditions:

* Patients with Chronic Kidney Disease previously evaluated by the nephrology service.
* History of requiring renal replacement therapy (hemodialysis, peritoneal dialysis, or kidney transplantation).
* Patients hospitalized within the last 3 months with a diagnosis of kidney failure.
* Patients with a known prior diagnosis of Autosomal Dominant Polycystic Kidney Disease or glomerular diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease who are referred to nephrology teleconsultation from primary care
Sampling Method: Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Appropriate referral to teleconsultation | Baseline
  Proportion of patients referred to nephrology teleconsultation during 2024 in a timely manner and with appropriate treatment. Timely referral is defined as referral within three months of the appearance of nephrology referral criteria. Treatment adequacy will be assessed based on the recommendations of the SEMERGEN Primary Care guidelines and the therapeutic harmonization protocols established by CatSalut.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Manzur, MD, Principal Investigator — CSAPG
Locations (1):
- Consorci Sanitari Alt Penedés-Garraf, Sant Pere de Ribes, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.